CLINICAL TRIAL: NCT05170165
Title: A Pilot Study to Increase Utilization of Guideline Directed Medical Therapy in Patients With HFrEF
Brief Title: A Pilot Study to Increase Utilization of GDMT in Patients With HFrEF
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Raj Khandwalla, Director of Cardiovascular Education, Cedars Sinai Care Foundation, Cedars-Sinai Medical Center
Other Study IDs: HFDTx study 1618
Record Dates: First submitted 2021-12-22; First posted 2021-12-27 (Actual); Last update posted 2023-09-05 (Actual); Status verified 2023-08

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Enrolled Subjects: Test a clinical decision support (CDS) tool that provides clinicians (cardiologists and nurse practitioners) recommendations regarding guideline directed medical therapy (GDMT) in patients with heart failure and reduced ejection fraction (HFrEF).
  Interventions: Other: Using a clinical decision software to provide specific recommendation of a medication at a certain dosage

INTERVENTIONS:
Other: Using a clinical decision software to provide specific recommendation of a medication at a certain dosage — During routine follow-up, clinicians, cardiologists, and NPs who have a scheduled visit with an enrolled patient will be offered a medication recommendation. The medication recommendation will be generated by the clinical decision support tool. The software will advise the cardiologist whether an HF medication should be initiated, discontinued, or the dosage titrated and if the patient requires labs. In addition, the software, or decision engine (DE), will be run once weekly and every time the patient has new basic metabolic panel results. If the patient is admitted to the hospital, skilled nursing facility, or inpatient rehabilitation unit, the use of DE will be placed on hold until the patient is discharged and at home.

SUMMARY:
The purpose of this study is to test a clinical decision support (CDS) tool that provides clinicians (cardiologists and nurse practitioners) medication recommendations regarding guideline directed medical therapy (GDMT) in patients with heart failure and reduced ejection fraction (HFrEF).

DETAILED DESCRIPTION:
The purpose of our study is to test whether home blood pressure monitoring (HBPM) with clinical-decision support (CDS) will optimize the use of GDMT in patients with HFrEF. HBPM allows cardiologists and NPs to monitor patients outside the clinical setting so that GDMT can be safely initiated and up-titrated. The CDS employs HBPM and electronic medical record (EMR) data to implement the ACC/AHA HF guidelines and provides cardiologists and NPs with GDMT recommendations.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of HFrEF (left ejection fraction < 40%, assessed by transthoracic echo, cardiac MRI, cardiac SPECT) within the past year.
* New York Heart Association (NYHA) class II-III at most recent screening assessment.
* GDMT composite score of less than or equal to 50% at baseline

Exclusion Criteria:

* Previous contraindication to beta blockers, ACE inhibitors, and/or ARB.
* Baseline creatinine > 2 mg/dl or potassium level at baseline > 5 mEq/L or eGFR <30 mL/min/1.73 m2.
* Baseline systolic blood pressure < 100 mmHg.
* Concomitant use of ACE, ARB, and/or ARNI
* Polycystic kidney disease
* History of angioedema
* History of or currently on a transplant list
* Left ventricular assist device
* Uncontrolled asthma
* Severe COPD
* Cirrhosis
* Currently receiving hospice or comfort care
* Patient not proficient with written and spoken English
* Patient has diminished decision making capability
* History of non-compliance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients >18 years with HFrEF who have suboptimal HF medical regimen
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-01-12 (Actual); Primary Completion 2023-09-25 (Estimated); Study Completion 2023-09-25 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients at or above 50% target dose of GDMT in HFrEF patients | 6 months
  Change in the proportion of patients at or above 50% target dose of GDMT in

SECONDARY OUTCOMES:
Percentage of accepted medication recommendations | 6 months
  The percentage of DE output medication recommendations in which the clinician accepts alerts

CONTACTS AND LOCATIONS:
Overall Officials: Raj Khandwalla, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars Sinai Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data that underlie the results after deidentification.
Supporting Information: Study Protocol, ICF
Time Frame: Immediately following publication and ending 2 years.
Access Criteria: Researchers who provide a methodologically sound proposal.